CLINICAL TRIAL: NCT04678440
Title: A Pilot Study of [18F]F-AraG Pharmacokinetics in Tumors and Non-Malignant Tissue Using Dynamic Total Body PET Imaging in Healthy Subjects and in Patients With Non-Small Cell Lung Cancer (NSCLC)
Brief Title: [18F]F-AraG/Total Body PET Imaging and Healthy Subjects and Lung Cancer Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: CellSight Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Simon R. Cherry, Professor, University of California, Davis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1630355; CST-FARAG-203 (Other: Cellsight)
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: total body positron emission tomography
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Healthy volunteers and patients with non-small cell lung cancer will undergo identical total-body PET scans. Lung cancer patients will undergo an additional PET scans after starting treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): Study participants will undergo a single dynamic [18F]F-AraG PET/CT scan (of duration up to 90-minutes) on the uEXPLORER PET/CT scanner. There will be a follow-up visit or call 7 days after the scan to assess any adverse events that could be attributed to either the scan or the administration of [18F]F-AraG.
  Interventions: Drug: [18F]F-AraG Imaging
- Non-Small Cell Lung Cancer Patients (NSCLC) (Experimental): Study participants with NSCLC who are planned to receive PD-1/PD-L1 immunotherapy will undergo a pre-therapy dynamic [18F]F-AraG PET/CT scan, and an optional post-therapy (first dose only) dynamic [18F]F-AraG PET/CT scan on the uEXPLORER total-body scanner.
  Interventions: Drug: [18F]F-AraG Imaging

INTERVENTIONS:
Drug: [18F]F-AraG Imaging — Total body PET imaging using [18F]F-AraG

SUMMARY:
In this pilot study, healthy volunteers and patients with Non-Small Cell Lung Cancer will undergo [18F]F-AraG dynamic imaging on the uEXPLORER total body Positron Emission Tomography/Computerized Tomography scanner to obtain preliminary data regarding pharmacokinetics and early biodistribution images.

DETAILED DESCRIPTION:
[18F]F-AraG, a fluorine-18 labeled analog of an FDA approved drug (Nelarabine) is a new imaging tracer targeted at imaging activated T-cells. Given that immunotherapeutic strategies, in particular immune checkpoint antibodies, focus on the generation of T-cell-based antitumor immunity, uptake of [18F]F-AraG within the tumor is hypothesized to correlate with T-cell mediated immune response seen in the biopsy samples of cancer patients treated with immune checkpoint blockade. Correlation of pre- and post-treatment intratumoral immune infiltration by means of PET imaging will guide the development of future clinical trials investigating the role of [18F]F-AraG in the monitoring of anti-tumor immune responses. Therefore, proper quantification of [18F]F-AraG uptake in tumor lesions, and understanding its relation with physiologic uptake in background tissues is important. Note: checkpoint therapy in this study is standard-of-care and is not under investigation.

Available PET/CT scanners can obtain dynamic images only on a portion of the body as large as their axial field of view, generally anywhere between 15-30 cm. The 194 cm long uEXPLORER total-body PET scanner is the world's first device to offer the ability to tomographically image all parts of the body simultaneously. Thus, the uEXPLORER PET/CT (now commercially available and with FDA 510(k) clearance) is the only scanner in the world capable of acquiring total-body dynamic images.

In this pilot study, 2-4 healthy volunteers will undergo [18F]F-AraG dynamic imaging on the uEXPLORER total body PET/CT scanner to obtain preliminary data regarding pharmacokinetics and early biodistribution images. In addition, 2-4 patients with NSCLC and planned for standard-of-care PD-1/PD-L1 immunotherapy will undergo [18F]F-AraG dynamic imaging similarly on the uEXPLORER total body PET/CT scanner to obtain data regarding pharmacokinetics of the tracer in tumor lesions in the context of normal tissue uptake. An optional second similar scan will be performed 7-14 days after the first dose of immunotherapy to explore and document any treatment related changes in [18F]F-AraG uptake and kinetics.

The study and data collected will be important to recommend an ideal time to acquire a whole body static scan using conventional and widely available PET/CT scanners for adequate tumor to background contrast and quantification, which in turn, will be essential for further clinical development of [18F]F-AraG to aid the monitoring of anti tumor immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Ability to understand the purposes and risks of the trial and has signed an IRB-approved informed consent form.
3. Willingness and ability to comply with all protocol required procedures.
4. For men and women of child-producing potential, willingness to use of effective double barrier contraceptive methods during the study, up to 1 day after the last administration of the investigational product.

   For NSCLC subjects only:
5. Patients with histologically confirmed advanced, locally advanced, or localized NSCLC.
6. Planned to undergo treatment with a PD-1 or PD-L1 inhibitor either as 1) monotherapy or as combination therapy with concurrent chemotherapy as treatment for advanced/metastatic disease; 2) As consolidation therapy following chemoradiation for locally advanced disease or 3) As induction therapy either as monotherapy or combination therapy with chemotherapy prior to planned surgical resection
7. At least 1 tumor lesion > 1 cm (cannot be only in liver) documented on CT or MRI or FDG-PET/CT (RECIST criteria 1.1; >1.5 cm for nodal lesions) within 45 days prior to scan date.
8. Per investigator's assessment and in consultation with oncologists, at least one eligible lesion must be sufficiently separated from tissues with known high [18F]F-AraG uptake, such as salivary glands, bladder, liver and kidneys so that quantification will be feasible.
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
10. Meeting all clinical safety lab values per institution's standard of care, or Investigator's discretion, for patients receiving cancer treatment.

Exclusion Criteria:

Subjects are not eligible if they meet ANY of the following criteria:

1. Serious comorbidities (nonmalignant disease or other conditions) that in the opinion of the investigator could compromise protocol objectives.
2. History of recent COVID-19 infection within the last 2 months OR history of COVID requiring hospitalization with lung injury at Investigator's discretion
3. Subjects with a diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the scan
4. Subjects receiving therapy with nucleoside analogs including but not limited to: acyclovir, valaclovir, penciclovir, famciclovir, ganciclovir, ribavirin, valganciclovir, glanciclovir
5. Pregnant women or nursing mothers.
6. Body weight more than 240 kg (529 pounds)

   For NSCLC subjects only:
7. Prior Treatment with anti-PD-1/PD-L1 immunotherapy.

   For Healthy subjects
8. No primary care physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon R Cherry, PhD, Principal Investigator — UC Davis
Locations (1):
- UC Davis EXPLORER Molecular Imaging Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-total-body-pet-imaging-study-in-healthy-subjects-and-lung-cancer-patients-372396/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteers | Non-Small Cell Lung Cancer Patients (NSCLC)
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Non-Small Cell Lung Cancer Patients (NSCLC) | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (46) | 53 (0) | 55 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Data on Whole-body Pharmacokinetics of [18F]F-AraG Physiologic Uptake in Various Healthy Tissues
Description: Data on [18F]F-AraG uptake in several tissue types will be collected from healthy subjects. This data will be presented in the form of time-activity curves (TAC) generated for each tissue type. Quantitative assessment of [18F]F-AraG biodistribution in healthy tissues will be reported as a function of time as mean Standard Uptake Value (SUV)
Time Frame: Baseline
Population: This outcome measure is only measured in the healthy subjects.
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 4
SUV
  Blood Pool | 0.31 (0.01)
  Myocardium | 4.36 (0.27)
  Brain | 0.04 (0.01)
  Kidney | 32.88 (5.42)
  Liver | 16.05 (2.03)
  Spleen | 3.46 (0.41)
  Muscle | 1.05 (0.26)
  Lungs | 0.67 (0.12)
  Bone Marrow | 1.46 (0.23)
  Lymph Nodes | 1.57 (0.51)

2. Primary Outcome: Data on Whole-body Pharmacokinetics of [18F]F-AraG Pathologic Uptake in Tumor Lesions Relative to Uptake in Background Tissues in NSCLC Subjects
Description: Data on [18F]F AraG uptake in tumor lesions and background activity in the same tissues as in Outcome 1 will be collected. This data will be similarly presented in the form of time-activity curves (TAC) generated for each tissue type, as well as for tumor lesions against their background tissues.
Time Frame: Baseline and 7-14 days after first dose of PD-1/PD-L1
Population: Mean and standard deviations are reported across seven different tumor sites and four different lymph nodes.
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Non-Small Cell Lung Cancer Patients (NSCLC)
Number analyzed (Participants) | 1
SUV
  Tumor (baseline) | 2.14 (0.20)
  Tumor (after therapy) | 2.30 (0.54)
  Mediastinal Lymph Nodes (Baseline) | 2.54 (0.69)
  Mediastinal Lymph Nodes (after therapy) | 3.15 (0.58)

3. Primary Outcome: Tumor-to-Background SUVR Over Time to Determine Earliest Adequate Uptake
Description: We will calculate the tumor-to-background Standardized Uptake Value Ratio (SUVR) at multiple time points. The primary aim is to identify the earliest time at which the SUVR indicates adequate tumor uptake relative to non-malignant tissue. This will guide recommendations for the ideal imaging start time for static whole-body scans.
Time Frame: Baseline and 7-14 days after first dose of PD-1/PD-L1
Measure: Mean (Standard Deviation); unit: SUV to blood ratio (SUVR)
Groups:
- Healthy Volunteers: Study participants will undergo a single dynamic [18F]F-AraG PET/CT scan (of duration up to 90-minutes) on the uEXPLORER PET/CT scanner.
  [18F]F-AraG Imaging: Total body PET imaging using [18F]F-AraG
- Non-Small Cell Lung Cancer Patients (NSCLC) - Pre-Therapy Scan: Study participants with NSCLC who are planned to receive PD-1/PD-L1 immunotherapy will undergo a pre-therapy dynamic [18F]F-AraG PET/CT scan, and an optional post-therapy (first dose only) dynamic [18F]F-AraG PET/CT scan on the uEXPLORER total-body scanner.
  [18F]F-AraG Imaging: Total body PET imaging using [18F]F-AraG
- Non-Small Cell Lung Cancer Patients (NSCLC) - 7 to 14 Days Post Therapy: Study participants with NSCLC who are planned to receive PD- 1/PD-L1 immunotherapy will undergo a pre-therapy dynamic [18F]F-AraG PET/CT scan, and an optional post-therapy (first dose only) dynamic [18F]F-AraG PET/CT scan on the EXPLORER total-body scanner.
  [18F]F-AraG Imaging: Total body PET imaging using [18F]F-AraG
Arm/Group | Healthy Volunteers | Non-Small Cell Lung Cancer Patients (NSCLC) - Pre-Therapy Scan | Non-Small Cell Lung Cancer Patients (NSCLC) - 7 to 14 Days Post Therapy
Number analyzed (Participants) | 4 | 1 | 1
SUV to blood ratio (SUVR)
  Myocardium | 13.72 (0.75) | 16.9 (NA) — Only 1 subject | 12.3 (NA) — Only 1 subject
  Brain | 0.13 (0.03) | 0.07 (NA) — Only 1 subject | 0.06 (NA) — Only 1 subject
  Kidney | 109.55 (28.88) | 133.0 (NA) — Only 1 subject | 150.2 (NA) — Only 1 subject
  Liver | 54.75 (12.38) | 76.5 (NA) — Only 1 subject | 67.4 (NA) — Only 1 subject
  Spleen | 11.60 (1.73) | 11.7 (NA) — Only 1 subject | 10.2 (NA) — Only 1 subject
  Muscle | 3.04 (0.20) | 3.93 (NA) — Only 1 subject | 1.90 (NA) — Only 1 subject
  Lungs | 1.83 (0.37) | 1.65 (NA) — Only 1 subject | 1.76 (NA) — Only 1 subject
  Bone Marrow | 4.87 (1.04) | 4.41 (NA) — Only 1 subject | 4.11 (NA) — Only 1 subject
  Mediastinal Lymph Nodes | 5.68 (1.33) | 8.59 (NA) — Only 1 subject | 9.50 (NA) — Only 1 subject
  Tumor | NA (NA) — No tumors in normal subjects | 4.79 (NA) — Only 1 subject | 6.02 (NA) — Only 1 subject

ADVERSE EVENTS:
Time Frame: Report initiation for all AEs and serious adverse events (SAEs) will begin immediately after the first infusion of [18F]F AraG (Visit 2) and continue until the Day 7 follow up.
Description: The definition of AE and SAE collection does not differ from the clinicaltrials.gov definition. There were no AEs or SAEs reported throughout the data collection timeline.
Arm/Group | Healthy Volunteers | Non-Small Cell Lung Cancer Patients (NSCLC)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/4 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT04678440/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT04678440/ICF_001.pdf